CLINICAL TRIAL: NCT04807205
Title: Post Market Study Using The Elite IQ Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN20-ELITEIQ-02
Record Dates: First submitted 2021-03-11; First posted 2021-03-19 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Hair Removal; Pseudo Folliculitis Barbae; Benign Vascular Lesion; Pigmented Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Elite IQ Laser (Experimental): The Elite IQ will be used on multiple areas of the body such as, but not limited to, the face, legs, and arms.
  Interventions: Device: RF Non-Invasive Treatment

INTERVENTIONS:
Device: RF Non-Invasive Treatment — Self-controlled single-arm group using the Elite IQ device

SUMMARY:
This is a prospective, open label, single-center clinical study to collect safety and efficacy data on the Elite iQ workstation. The intended use of the Elite iQ device used in this study is for the treatment of hair removal, pseudo folliculitis barbae, and benign vascular and pigmented lesions.

DETAILED DESCRIPTION:
Up to 20 subjects will be enrolled at up to 1 study center. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 5 treatments on multiple areas of the body such as, but not limited to, the face, legs, and arms. All subjects will be required to return a follow-up visit at 30 - 90 days after the final treatment in each treatment area.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 years of age or older.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* The subject is hypersensitive to light in the near infrared wavelength region
* The subject has sun-damaged skin (treatment contraindicated with Alex laser only)
* The subject had recent unprotected sun exposure (for Alex laser within four weeks of treatment; for Nd:YAG laser within one week of treatment), including the use of tanning beds or tanning products, such as creams, lotions and sprays
* The subject is taking medication which is known to increase sensitivity to sunlight
* The subject has seizure disorders triggered by light
* The subject is taking anticoagulants
* The subject is taking or have taken oral isotretinoin, such as Accutane®, within the last six months
* The subject is taking medication that alters the wound-healing response
* The subject has a history of healing problems or history of keloid formation
* The subject has an active localized or systemic infection, or an open wound in area being treated
* The subject has a significant systemic illness or an illness localized in area being treated
* The subject has a history of skin cancer or suspicious lesions
* The subject has an autoimmune disease
* The subject is receiving or have received gold therapy
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months to entering this study.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (1):
- Scripps Clinic Carmel Valley, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Elite IQ Laser
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elite IQ Laser
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14
  Hispanic | 3
  Asian | 2
  African American | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants]
  Fitzpatrick Skin Type I | 0
  Fitzpatrick Skin Type II | 7
  Fitzpatrick Skin Type III | 8
  Fitzpatrick Skin Type IV | 2
  Fitzpatrick Skin Type V | 2
  Fitzpatrick Skin Type VI | 1

OUTCOME MEASURES:

1. Primary Outcome: Blinded Evaluation of Pre-treatment Images vs. Follow up Images to Determine Which Image Was Taken Pre-treatment vs. at the Follow up.
Description: Blind identification of pre-treatment images vs. 60 day follow up images. It is performed by independent reviewers. The outcome will be reported as a percentage of photographs identified correctly.
Time Frame: 60 day (+/- 30 days) post last treatment
Population: Three subjects had an extra treatment area treated, and were graded for each separate treatment area, so the total number of treatment areas graded was 23 (23 photos were analyzed). Each photo was graded by 3 individual graders, for a total of 69 photos being analyzed. The average percentage of photographs identified correctly of these 3 graders is reported.
Measure: Mean (Standard Deviation); unit: % of photos correctly identified
Units Other Than Participants: Photos
Arm/Group | Elite IQ Laser
Number analyzed (Participants) | 20
Number analyzed (Photos) | 69
% of photos correctly identified | 94.2 (.05)

2. Secondary Outcome: Principle Investigator Assessment Using the Global Aesthetic Improvement Scale (PGAIS)
Description: Principle Investigator assessment using the Global Aesthetic Improvement Scale (PGAIS) at the 60 day follow up visit. The GAIS scale ranges from 1 to 5, with 1 being "very much improved," 2 being "much improved," 3 being "improved," 4 being "no change," and 5 being "worse." This is the count of the number of subjects who the physician graded a 3 or higher.
Time Frame: 60 day (+/- 30 days) post last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Elite IQ Laser
Number analyzed (Participants) | 20
Participants | 20

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction rates at the 60 day follow up visit. The subject satisfaction scale ranges from 1 to 6, with 1 being extremely unsatisfied, 2 being dissatisfied, 3 being slightly unsatisfied, 4 being slightly satisfied, 5 being satisfied, and 6 being extremely satisfied. This is the count of the number of subjects who graded themselves a 4 or higher.
Time Frame: 60 day (+/- 30 days) post last treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Elite IQ Laser
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: All adverse events were collected and resolved during the time period of when the study started to the final follow up date (6 months post last treatment, up to a total of 9 months)
Arm/Group | Elite IQ Laser
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elite IQ Laser (N=20)
Blistering (Skin and subcutaneous tissue disorders) | 2
Crusting (Skin and subcutaneous tissue disorders) | 4
Edema (Skin and subcutaneous tissue disorders) | 20
Erythema (Skin and subcutaneous tissue disorders) | 20
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT04807205/Prot_SAP_001.pdf